CLINICAL TRIAL: NCT05221346
Title: Effect of Oleactiv® on LDL Oxidability in Volunteers With Moderate Hypercholesterolemia - a Controlled, Randomized, Double-blind Study
Brief Title: Effect of Oleactiv® on LDL Oxidability
Acronym: e-POL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Principal investigator, Institut Pasteur de Lille
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-A00508-33
Record Dates: First submitted 2022-01-07; First posted 2022-02-03 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Hypercholesterolemia
Keywords: Polyphenols; LDL oxidability
MeSH Terms: conditions — Hypercholesterolemia | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant food supplement (Experimental): * Dietary supplements in capsule form
  * 1 capsule per day at breakfast
  Interventions: Dietary Supplement: Plant food supplement
- Maltodextrin (Placebo Comparator): * Dietary supplements in capsule form
  * 1 capsule per day at breakfast
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Plant food supplement — Food supplements are consumed during 3 weeks by hypercholesterolemic volunteers
  Arms: Plant food supplement
Dietary Supplement: Maltodextrin — Food supplements are consumed during 3 weeks by hypercholesterolemic volunteers
  Arms: Maltodextrin

SUMMARY:
Oleactiv® have previously demonstrated beneficial effects in an animal model of diet-induced atherosclerosis. After a 12-week supplementation, a substantial reduction of aortic fatty streak area has been observed. Also, Oleactiv®-supplemented hamsters displayed significant decrease of both non-HDL-cholesterol and triglycerides levels. Also, phenolic compounds from Oleactiv® demonstrated that increase of cholesterol efflux capacity (CEC) is one of the mechanisms that may explain preventive effect on atheroma development.

These effects observed in animals will thus be investigated in human. The main hypothesis of the present study is that phenolic compounds from Oleactiv® may improve LDL oxidability in volunteers with moderate hypercholesterolemia after 3 weeks of consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male aged between 40 and 70 years (limits included),
* BMI between 20 and 30 kg / m² (limits included)
* Weight over 65kg (to respect volume blood collection reglementation)
* Fasting plasma LDL cholesterol between 1.16 g / L and 1.9 g / L (limits included) if the cardiovascular risk is low OR Fasting plasma LDL cholesterol between 1.0 g / L and 1.9 g / L (limits included) if the cardiovascular risk is moderate (SCORE calculated according to the European Society of Cardiology 2019)
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme.

Exclusion Criteria:

* Dyslipidemia or hyperlipidemia:

  * Fasting total cholesterol ≥ 3.0 g / L
  * Fasting triglycerides> 2 g / L
  * with heterozygous familial hypercholesterolemia
* Hypertensive-treated
* Diabetes treated or not with medication
* Taking drugs known to have an impact on lipid metabolism (statin, ezetimibe, colestyramine, fibrate, etc.) in the month preceding inclusion and / or likely to consume them during the test
* Consuming food supplements or functional foods known to have an influence on cholesterolemia (phytosterol, phytostanol, red rice yeast, policosanols, beta-glucans at a dose greater than 3 g / d) in the month preceding the inclusion and / or likely to take during the test
* Consuming probiotics in the form of a food supplement in the month preceding inclusion and / or likely to take them during the test
* Following or having followed a hypocaloric diet (energy intake <1,500 kCal / day) in the month preceding inclusion and / or likely to undertake this diet during the test
* Who donated blood in the 3 months preceding inclusion
* Diagnosed eating disorders (bulimia, anorexia nervosa, vomiting)
* High level athlete (physical activity for 1 hour per day)
* Smoking more than 5 cigarettes per day
* Bariatric surgery or who has a gastroplasty ring
* Consuming more than 3 standard drinks of alcoholic beverage daily,
* Consuming drugs,
* Suffering from serious illnesses such as cancer, recent myocardial infarction, serious digestive pathologies or others diseases found to be inconsistent with the conduct of the study by the investigator,
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Any other condition which in the investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.
* Known allergy to one of the component of the supplement (Grape, olive, artichoke, blackcurrant or pomegranate) or to corn.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of LDL oxidability after 3 weeks of food supplement consumption compared to placebo group | 3 months
  LDL oxidability

SECONDARY OUTCOMES:
Change from baseline of lipid metabolism after 3 weeks of food supplement consumption compared to placebo group | 3 months
  Total cholesterol, HDL, LDL, Triglycerides,
Change from baseline of lipoproteins size distribution after 3 weeks of food supplement consumption compared to placebo group | 3 months
  Lipoprotein size
Change from baseline of plasma paraoxonase activity after 3 weeks of food supplement consumption compared to placebo group | 3 months
  Paraoxonase activity
Change from baseline of reverse transport of cholesterol after 3 weeks of food supplement consumption compared to placebo group | 3 months
  Reverse transport of cholesterol
Change from baseline of cholesterol load capacity after 3 weeks of food supplement consumption compared to placebo group | 3 months
  Cholesterol load capacity
Maximum plasma concentration of phenolic compounds in a 24h-blood collection | 3 months
  Phenolic compounds were measured after food supplement consumption at 7 points (T0, T1h, T2h, T4h, T6h, T10h, T24h).
Time of complete elimination of phenolic compounds in a 24h-blood collection | 3 months
  Phenolic compounds were measured after food supplement consumption at 7 points (T0, T1h, T2h, T4h, T6h, T10h, T24h).
Maximum plasma concentration of oxidized LDL in a 24h-blood collection | 3 months
  Oxidized LDL were measured after food supplement consumption at 7 points (T0, T1h, T2h, T4h, T6h, T10h, T24h).
Maximum concentration of urinary isoprostanes in a 48h-urine collection | 3 months
  Urinary isoprostanes were measured after food supplement consumption at 7 points (from 22h the day before to 8h (T0), T0-6h, T6-10h, T10-14h, T14-24h, T24-32h, T32-48h).
Change from baseline of carbohydrate metabolism after 3 weeks of food supplement consumption compared to placebo group | 3 months
  glycemia, insulin
Change from baseline of arterial stiffness after 3 weeks of food supplement consumption compared to placebo group | 3 months
  Arterial stiffness via the Sphygmocor® measuring device

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Lecerf, MD, Principal Investigator — Institut Pasteur de Lille - NutrInvest
Locations (1):
- NutrINvest, Lille, France

IPD SHARING:
Plan to Share IPD: No
IPD will available only for sponsor